CLINICAL TRIAL: NCT03140761
Title: The Prevalence of Secondary Adrenal Insufficiency in Patients With Exacerbation of COPD in Glucocorticoid Treatment Related to Differenct Gene Polymorphisms of the Glucocorticoid Receptor Gene
Status: Completed | Type: Observational
Sponsor: Chronic Obstructive Pulmonary Disease Trial Network, Denmark (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Pradeesh Sivapalan, MD, Phd fellow, Chronic Obstructive Pulmonary Disease Trial Network, Denmark
Other Study IDs: COPTRIN
Record Dates: First submitted 2017-04-17; First posted 2017-05-04 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Adrenal Insufficiency
MeSH Terms: conditions — Adrenal Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — Blood samples and DNA from gene analyses
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate the correlation between four well-known polymorphisms of the glucocorticoid receptor gene (two with reduced sensitivity versus two with increased sensitivity) and the prevalence of secondary adrenal insufficiency in glucocorticoid-treated patients with exacerbation of COPD.

DETAILED DESCRIPTION:
COPD patients who have received systemic glucocorticoid exceeding the equivalent of 180 mg prednisolone which are homo / heterozygous for the BclI and / or N363S polymorphisms (associated with increased glucocorticoid sensitivity) will have a lower cortisol response in a synacthen® test (greater suppression of adrenal corticosteroid) than the corresponding patients there are wild-type or homo- or heterozygous for the polymorphic ER22 / 23EK and / or 9β (associated with decreased sensitivity). Information from the results of the investigation will be able to help clinicians to identify patients with acute exacerbation of COPD (AECOPD) at risk of of secondary adrenal insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients > 18 years
* Caucasian classified with COPD
* Patients with AECOPD being treated with at least 5 days of glucocorticoid (minimum of 180 mg)

Exclusion Criteria:

* Treated with estrogen-containing medications, including anticonceptiva 6 weeks prior to Synacthen®
* Pregnancy or lactation
* on regular systemic glucocorticoid therapy before admission to the hospital
* People who are detained under the act on the use of coercion in psychiatry
* Severe language problems or inability to provide written informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 78 hospitalised patients with exacerbation of COPD
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-05-09 (Actual)

PRIMARY OUTCOMES:
Secondary Adrenal insufficiency | average 1 month
  test for adrenal function by stimulation test

SECONDARY OUTCOMES:
Metabolic syndrome | average 1 month
  blood lipids, blood pressure, plasma glucose, abdominal obesity, body composition
Bone mineral loss | average 1 month
  bonemarkers
Onset of Diabetes Mellitus | average 1 month
Quality of life | average 1 month
  test by questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal medicine, Herlev & Gentofte Universtity Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Undecided